CLINICAL TRIAL: NCT01789905
Title: Tygacil Drug Use Investigation (Tigecycline Evaluation Study For Safety And Effectiveness In Patient Infected With Multi-Drug Resistance.)
Brief Title: Tygacil Drug Use Investigation
Acronym: TIGER
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1811187
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Intra-Abdominal Infections; Skin Disease, Infectious
Keywords: Tygacil; Tigecycline; Post marketing surveillance; Japanese; Infection
MeSH Terms: conditions — Intraabdominal Infections; Skin Diseases, Infectious; Infections | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tigecycline (Tygacil): Subjects who are treated with tigecycline
  Interventions: Drug: Tigecycline (Tygacil)

INTERVENTIONS:
Drug: Tigecycline (Tygacil) — Tigecycline 50 mg intravenously. Therapy conducted according to Japanese LPD of Tygacil. Tygacil will be dosed according to labeling. The administration and duration of the therapy will be determined by the treating physician to meet the patient individual needs for treatment.
  Other Names: Tygacil, Tigecycline

SUMMARY:
Secondary Data Collection Study; safety and effectiveness of Tigecycline .under Japanese medical practice

ELIGIBILITY:
Inclusion Criteria:

* All patients who are prescribed tigecycline (Tygacil).

Exclusion Criteria:

* Subject who have not been prescribed tigecycline (Tygacil).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving B1811187 prescribes the tigecycline (Tygacil).
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2013-04-15 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1811187&StudyName=Tygacil%20Drug%20Use%20Investigation

RESULTS

PARTICIPANT FLOW:
Groups:
- Tygacil (Tigecycline): Participants who received Tygacil as indicated in the approved local product document were observed for a period of 14 days at maximum. The follow-up period was 28 days post-treatment. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Tygacil (Tigecycline)
Started | 116
Completed | 116
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 116 participants were registered in this study. There was no participant excluded from the baseline analysis.
Arm/Group | Tygacil (Tigecycline)
Number analyzed (Participants) | 116
Age, Customized [Number; unit: Participants]
  <15 years | 5
  ≥15 and <65 years | 47
  ≥65 years | 64
Sex/Gender, Customized [Number; unit: Participants]
  Male | 64
  Female | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reaction (ADR)
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Tygacil in a participant who received Tygacil. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Tygacil was assessed by the physician.
Time Frame: Up until 14 days from the start date and 28 days from the end of the observation period
Population: The safety analysis set comprised of participants who had received Tygacil at least once.
Measure: Number; unit: Participants
Arm/Group | Tygacil (Tigecycline)
Number analyzed (Participants) | 116
Participants
  ADR | 41
  Serious ADR | 15

2. Secondary Outcome: Clinical Response Rate
Description: Clinical response rate, which was defined as the percentage of participants who achieved clinical response as "effective" over the total number of assessable effectiveness analysis population("effective" plus "ineffective",) was presented along with two-sided 95% CI. Clinical response of Tygacil was assessed as "effective," "ineffective," or "indeterminate" by the physician at the end of observation period. Overall response of Tygacil was determined by the physician based on laboratory and clinical findings without bacteriological findings.
Time Frame: Within 14 days from the start date
Population: The analysis set comprised of participants in the safety analysis set who had effectiveness evaluation at the end date of the observation period at least once. Participants evaluated as "indeterminate (n=28)" were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tygacil (Tigecycline)
Number analyzed (Participants) | 116
Percentage of Participants | 73.9 [63.4 to 82.7]

3. Secondary Outcome: Clinical Response Rate of Cure
Description: The cure rate, which was defined as the percentage of participants who were assessed as "cure" over the total number of assessable effectiveness analysis population ("cure" plus "failure"), was presented along with two-sided 95% CI. Clinical response of cure was assessed as "cure," "failure," or "indeterminate" by the physician within 28 days post-treatment.
Time Frame: Within 28 days post-treatment
Population: The analysis set comprised of participants in the safety analysis set who had effectiveness evaluation at the Test-of-Cure visit at least once. Participants evaluated as "indeterminate (n=38) " were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tygacil (Tigecycline)
Number analyzed (Participants) | 116
Percentage of Participants | 59.0 [47.3 to 70.0]

ADVERSE EVENTS:
Time Frame: Up until 14 days from the start date and 28 days from the end of the observation period
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both serious and non-serious events during the study.
Arm/Group | Tygacil (Tigecycline)
All-Cause Mortality (participants affected / at risk) | 42/116
Serious Adverse Events (participants affected / at risk) | 49/116
Other Adverse Events (participants affected / at risk) | 54/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil (Tigecycline) (N=116)
Hypotension (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Renal impairment (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 2
Substance-induced psychotic disorder (Psychiatric disorders) | 1
Seizure (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Brain stem haemorrhage (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Platelet count decreased (Investigations) | 2
Hepatic enzyme increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Arterial injury (Injury, poisoning and procedural complications) | 1
Systemic candida (Infections and infestations) | 2
Superinfection (Infections and infestations) | 1
Stenotrophomonas infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 5
Sepsis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 5
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 2
Pathogen resistance (Infections and infestations) | 1
Oral viral infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Mucormycosis (Infections and infestations) | 1
Meningoencephalitis herpetic (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Encephalitis viral (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Cytomegalovirus enterocolitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Abdominal abscess (Infections and infestations) | 1
Graft versus host disease (Immune system disorders) | 1
Engraftment syndrome (Immune system disorders) | 1
Acute graft versus host disease (Immune system disorders) | 2
Venoocclusive liver disease (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 2
Pyrexia (General disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 6
Mucous membrane disorder (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Disease progression (General disorders) | 1
Condition aggravated (General disorders) | 7
Chest discomfort (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Eye pain (Eye disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Pancytopenia (Blood and lymphatic system disorders) | 2
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 4
Cytopenia (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil (Tigecycline) (N=116)
Decreased appetite (Metabolism and nutrition disorders) | 3
Delirium (Psychiatric disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 4
Hepatobiliary disease (Hepatobiliary disorders) | 3
Liver disorder (Hepatobiliary disorders) | 4
Renal impairment (Renal and urinary disorders) | 6
Blood alkaline phosphatase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 3
Pancreatic enzymes increased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT01789905/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT01789905/SAP_001.pdf